CLINICAL TRIAL: NCT02631733
Title: A Phase I Study of a Combination of MM-398 and Veliparib in Solid Tumors
Brief Title: Liposomal Irinotecan and Veliparib in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02125; NCI-2015-02125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-C-0012; 9914 (Other: Yale University Cancer Center LAO); 9914 (Other: CTEP); ZIABC011078 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2015-12-16 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Ferrosoferric Oxide; irinotecan sucrosofate; Magnetic Resonance Spectroscopy; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (liposomal irinotecan, veliparib) (Experimental): Patients receive liposomal irinotecan IV over 90 minutes on days 1 and 15 and veliparib PO BID on days 5-12 and 19-25 or 3-12 and 17-25. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Within 2-6 days prior to beginning liposomal irinotecan treatment, patients may optionally receive FMX IV and undergo MRI at baseline and 24 hours after FMX infusion.
  Interventions: Drug: Ferumoxytol; Drug: Irinotecan Sucrosofate; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Veliparib

INTERVENTIONS:
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Drug: Irinotecan Sucrosofate — Given IV
  Other Names: inotecan Hydrochloride as Sucrosulfate Salt Form Liposomal Formulation; Irinotecan Liposome; Irinotecan Sucrosofate Liposome; Irinotecan Sucrosofate-containing Pegylated Liposomal Formulation; MM 398; MM-398; MM398; nal-IRI; Nanoliposomal Irinotecan; Nanoliposomal Irinotecan as Sucrosofate; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP 02; PEP-02; PEP02
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with liposomal irinotecan in treating patients with solid tumors. Liposomal irinotecan and veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of escalating doses of liposomal irinotecan (MM-398) + veliparib combination.

II. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of MM-398 + veliparib.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To characterize the preliminary efficacy of the combination using key efficacy indicators, such as objective response rate, clinical benefit rate defined as complete response (CR), partial response (PR), or stable disease (SD) at 24 weeks, and progression free survival (PFS).

EXPLORATORY OBJECTIVE:

I. Imaging, tumor, and blood biomarkers to assess the sensitivity or resistance to each drug and/or correlation with clinical response.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive liposomal irinotecan intravenously (IV) over 90 minutes on days 1 and 15 and veliparib orally (PO) twice daily (BID) on days 5-12 and 19-25 or 3-12 and 17-25. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Within 2-6 days prior to beginning liposomal irinotecan treatment, patients may optionally receive ferumoxytol (FMX) IV and undergo magnetic resonance imaging (MRI) at baseline and 24 hours after FMX infusion.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed diagnosis of a solid tumor cancer for which there is no known standard therapy capable of extending life expectancy
* Prior poly ADP ribose polymerase (PARP) inhibitor therapy is allowed; patients with ovarian cancer and a BRCA mutation should have had prior treatment with olaparib per guidelines for standard of care treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Age >= 18 years
* Because no dosing or adverse event data are currently available on the use of veliparib in combination with MM-398 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Hemoglobin >= 10 g/dL (within 28 days prior to administration of ABT-888)
* Leukocytes >= 3,000/mcL (within 28 days prior to administration of ABT-888)
* Absolute neutrophil count >= 1,500/mcL without the use of hematopoietic growth factors (within 28 days prior to administration of ABT-888)
* Platelets >= 100,000/mcL (within 28 days prior to administration of ABT-888)
* Total bilirubin below institutional upper limit of normal (ULN) (within 28 days prior to administration of ABT-888)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (=< 5 x ULN is acceptable if liver metastases are present) (within 28 days prior to administration of ABT-888)
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (within 28 days prior to administration of ABT-888)
* Based on animal data, MM-398 (ONIVYDETM) and veliparib causes embryo toxicity and teratogenicity; thus, women of childbearing potential and male patients should use effective contraception during treatment with MM-398 and for 90 days following the final dose of veliparib and MM-398 for both female and male patients; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* IMAGING CORRELATIVE STUDY: Patients will be eligible to participate in the FMX imaging study if the participating study center offers this test and they do not meet any of the following criteria:

  * Evidence of iron overload as determined by:

    * Fasting transferrin saturation of > 45% and/or
    * Serum ferritin levels > 1000 ng/ml
  * A history of allergic reactions to any of the following:

    * Compounds similar to ferumoxytol or any of its components as described in full prescribing information for ferumoxytol injection
    * Any IV iron replacement product (e.g. parenteral iron, dextran, iron-dextran, or parenteral iron polysaccharide preparations)
    * Multiple drugs
  * Unable to undergo MRI or for whom MRI is otherwise contraindicated (e.g. presence of errant metal, cardiac pacemakers, pain pumps or other MRI incompatible devices; or history claustrophobia or anxiety related to undergoing MRI)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those whose adverse events have not resolved to grade 1 or less (except alopecia) from agents administered more than 4 weeks earlier; patients must have completed prior biological therapies and/or targeted therapies >= 2 weeks prior to study enrollment; patients who have had radiation to the pelvis or other bone marrow-bearing sites will be considered on a case by case basis and may be excluded if the bone marrow reserve is not considered adequate (i.e. radiation to > 25% of bone marrow)
* Patients who are receiving any other investigational agents
* Subjects with symptomatic brain metastases will be excluded from trial secondary to poor prognosis; however, subjects who have had treatment for their brain metastasis and whose brain disease is stable without steroid therapy for at least 3 months may be enrolled
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib and MM-398; if patients have a history of allergic reactions to compounds resembling MM-398, they will be excluded from participating in the FMX MRI study, if applicable
* Patients who have severe hypersensitivity to irinotecan hydrochloride (HCl)
* Patients with known and confirmed diagnosis of interstitial lung disease (IDL)
* Clinically significant gastrointestinal (GI) disorders, including history of small bowel obstruction unless the obstruction was a surgically treated remote episode
* Patient is unable to swallow or keep down oral medication
* Patients at the National Cancer Institute (NCI) site and other selected centers who are willing to undergo an optional pre-treatment ferumoxytol MRI must not have evidence of iron overload, a known hypersensitivity to ferumoxytol or any other IV iron product, a documented history of multiple drug allergies, or those for whom MRI is otherwise contraindicated, including claustrophobia or anxiety related to undergoing MRI; this exclusion criterion applies only to patients enrolling at NCI and other selected sites; of note, the principal investigator (PI) will allow other centers to offer FMX MRI scans if the site in question is willing and the site PI can identify the necessary resources and expertise at their center
* Active infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because veliparib, MM-398 and ferumoxytol are agents with the potential for teratogenic or abortifacient effects; because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with veliparib, MM-398 and/or ferumoxytol breastfeeding should be discontinued if the mother is treated with any of these agents; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with veliparib, MM-398 and/or ferumoxytol; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients who need chronic use of medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible
* Veliparib has a potential seizure risk, therefore patients with a high risk of seizures should be excluded from the protocol (e.g. those patients with an uncontrolled seizure disorder, and/or patients who have had a focal or generalized seizure within the last 12 months
* Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/myelodysplastic syndrome (MDS) or with features suggestive of AML/MDS
* Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 4 weeks
  Will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 as of April 1, 2018). Safety and tolerability of escalating doses of liposomal irinotecan and veliparib combination will be evaluated.
Maximum tolerated dose and recommended phase II dose of liposomal irinotecan in combination with veliparib | At 28 days
  Maximum tolerated dose and recommended phase II dose of liposomal irinotecan in combination with veliparib will be determined by incidence of dose limiting toxicities, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 as of April 1, 2018).

SECONDARY OUTCOMES:
Tumor response | Up to 4 weeks after completion of study treatment
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors version 1.1.
Objective response rate | At 24 weeks
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors version 1.1.
Clinical benefit rate defined as complete response, partial response, or stable disease | At 24 weeks
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors version 1.1.
Progression free survival | Duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up to 4 weeks after completion of study treatment
  Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

OTHER OUTCOMES:
Biomarker levels | Up to 4 weeks after completion of study treatment
  Will be studied to assess the sensitivity or resistance to each drug and correlated with clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, Principal Investigator — Yale University Cancer Center LAO
Locations (6):
- United States (6):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] LaRose M, Connolly RM, O'Sullivan CC, Velcheti V, Vilimas R, Gano K, Bates SE, Pommier Y, Thomas A. A Phase I Study of a Combination of Liposomal Irinotecan and Veliparib in Solid Tumors. Oncologist. 2023 May 8;28(5):460-e298. doi: 10.1093/oncolo/oyad023. PMID 37010988